CLINICAL TRIAL: NCT00194623
Title: Botox (Botulinum Toxin A) as a Treatment for Chronic Male Pelvic Pain Syndrome: A Randomized Placebo Controlled Trial
Brief Title: Botox as a Treatment for Chronic Male Pelvic Pain Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Reorganization of personnel forced termination.
Sponsor: University of Washington (Other)
Collaborators: Paul G. Allen Family Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 02-5458-A 04
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Chronic Male Pelvic Pain Syndrome
Keywords: prostatitis
MeSH Terms: conditions — Prostatitis | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botulinum Toxin A (Botox)

SUMMARY:
Chronic pelvic pain syndrome (CPPS) is thought to affect approximately 8% of men aged 18 and older. Patients with this condition experience pain in the perineum, the genitalia, and the rectum. As well, there is associated voiding, sexual, and ejaculatory dysfunction. The impact of patient well-being is thought to be equivalent to patients with congestive heart failure. The etiology of this condition is unknown, thus making treatment very difficult. Researchers have pursued an infectious cause for the disease; however, studies have failed to substantiate this theory. Despite this, the main treatment offered to patients is long-term antibiotic therapy. Results from this treatment modality have been unsatisfactory.

Other groups have postulated that the symptoms of CPPS may be secondary to neuromuscular factors. Some studies have demonstrated increases in pelvic muscular tone. Maneuvers such as prostate massage and levator massage have shown some benefit in relieving symptoms. Treatment with alpha-blockers to relax prostate smooth muscle has brought about improvement in a portion of patients. Use of generalized muscle relaxants has produced mediocre results.

However, many of these neuromuscular treatments are generalized and do not target the perineal musculature directly. It is theorized that spasm of the perineal muscles triggered by an unknown noxious stimuli (e.g. infection) cause the pain and symptoms of CPPS. At our center, we have performed pilot studies using botulinum toxin A. Four patients were treated with Botox". 100 U were injected in three locations in the midline of the bulbocavernosus muscle. The bulbocavernosus muscle is easily accessible and shares innervation with the pelvic musculature. Patient's response to medication was measured by the NIH Prostatitis pain scale and as well as the University of Washington prostatitis pain scale. All patients reported resolution of symptoms. Remission lasted for duration of 10-12 weeks. No patients reported adverse events.

HYPOTHESIS

Botulinum toxin A is effective in the treatment of chronic pelvic pain syndrome in men.

DETAILED DESCRIPTION:
Visit 1 Patient will review and sign the study consent form. Subject will be asked to complete questionnaires. Then, patient will then be asked to give a semen sample.

Visit 2 (1 week after Visit I) Prior to this visit, the patient will be randomized to either active medication or placebo. First, the patient will then undergo a physical exam including a genital and rectal exam. Then, the patient will be brought in to the room and placed in lithotomy position. The perineum will be prepped with iodine solution. EMG electrodes and a ground will be placed in the perineum. Three landmarks (1. middle of bulbospongiosus muscle; 2. perineal body; 3. an area equidistant from 1 and 2) will be marked using a skin marker. The EMG needle will be placed into each landmark and the patient will be asked to squeeze his perineal muscles. Once in the proper location, 1.3 cc of medication (active drug or placebo) will be distributed into these landmarks. The remaining 2.6 ccs will be injected into 2 other painful pelvic muscle sites as determined physical exam. The area will then be gently massaged.

1. Month Post Injection Mailing:

   The patient will be mailed a packet containing follow-up questionnaires.
2. Month Post Injection Mailing: Same as 1 Month Post Injection Visit.
3. Month Post Visit (Visit 3) First, the subject will be asked to fill out follow-up questionnaires. Next, a physical exam and prostate massage will be performed and expressed prostatic secretions collected. Finally, the subject will be asked to provide a semen sample.

Optional open label trial for those patients randomized to placebo section:

Open label injection visit (Visit 4) Injection of open label Botox as in Visit 2.

1. Month Post Open Label Botox Injection Mailing:

   The patient will be mailed a packet containing follow-up questionnaires.
2. Month Post Open Label Botox Injection Mailing:

   Same as 1 Month Post Injection mailing.
3. Month Post Open Label Injection Visit:

Same as Visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 and older
* History of chronic pelvic pain syndrome (NIH type IIIA and IIIB) for at least 3 months
* No antibiotics or new treatment for prostatitis for at least 30 days
* Written informed consent and written authorization for use or release of health and research study information have been obtained.
* Subject has severity/stage of disease: pain areas must include perineum.
* Laboratory findings required : negative urine cultures.
* Ability to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

* Documented urinary tract infection
* Bacteria isolated to the prostate from segmental urine cultures
* Pain from another source in the genitourinary tract (e.g. renal colic)
* Genitourinary (GU) malignancy
* History of radiation to the GU tract
* Previous or current botulinum therapy
* Known allergy or sensitivity to any study medication (Botox, lidocaine)
* Diagnosis of myasthenia gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis, spinal cord injury or any other significant disease which might interfere with neuromuscular transmission
* Concurrent use of aminoglycoside antibiotics or agents that interfere with neuromuscular transmission
* Profound atrophy or excessive weakness of the muscles to be injected
* Infection at the injection site or systemic infection
* Concurrent participation in another investigational drug study
* Is overtly psychotic or suicidal.
* Has post-surgical pain
* Has back or rectal pain only.
* Was treated for prostate, bladder, renal or other genitourinary malignancy
* Had in the past or is currently undergoing radiation therapy
* Has a history of genitourinary tuberculosis
* Is currently taking antibiotics.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-08; Study Completion 2007-08

PRIMARY OUTCOMES:
NIH-CPSI -pain scores at 3 months post-treatment follow-up | 3 months post treatment

SECONDARY OUTCOMES:
AUA score at 3 months post-treatment follow-up | 3 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Berger, MD, Principal Investigator — Professor of Urology